CLINICAL TRIAL: NCT01191723
Title: A Randomized, Double Blind, Placebo Controlled, Three- Period Crossover Study Comparing the Acute Effects of Orally Inhaled Dihydroergotamine (DHE), Oral Moxifloxacin, and Placebo on QT Intervals in Healthy Adults
Brief Title: QT Intervals Study to Compare the Acute Effects of Orally Inhaled Dihydroergotamine (DHE), Oral Moxifloxacin, and Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP0004-CL-P103
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A, then Treatment B, then Treatment C (Other): There was 48 hour wash-out between treatment visits. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 2.
  Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 3. Treatment C = inhaler placebo and placebo capsules at Visit 4. Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule
- Treatment A, then Treatment C, then Treatment B (Other): There was 48 hour wash-out between treatment visits. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 2.
  Treatment C = inhaler placebo and placebo capsules at Visit 3. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 4. Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule
- Treatment B, then Treatment A, then Treatment C (Other): There was 48 hour wash-out between treatment visits. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 2. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 3.
  Treatment C = inhaler placebo and placebo capsules at Visit 4. Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule
- Treatment B, then Treatment C, then Treatment A (Other): There was 48 hour wash-out between treatment visits. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 2. Treatment C = inhaler placebo and placebo capsules at Visit 3. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 4.
  Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule
- Treatment C, then Treatment A, then Treatment B (Other): There was 48 hour wash-out between treatment visits. Treatment C = inhaler placebo and placebo capsules at Visit 2. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 3.
  Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 4. Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule
- Treatment C, then Treatment B, then Treatment A (Other): There was 48 hour wash-out between treatment visits.
  Treatment C = inhaler placebo and placebo capsules at Visit 2. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 3. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 4.
  Tablets were orally administered after oral inhalation dosing.
  Interventions: Drug: MAP0004; Drug: Inhaler Placebo; Drug: Moxifloxacin; Drug: Placebo Capsule

INTERVENTIONS:
Drug: MAP0004 — 3.0mg orally inhaled MAP0004 administered in Treatment B as per protocol
Drug: Inhaler Placebo — Placebo for Inhaler administered in Treatments A and C
Drug: Moxifloxacin — 400mg encapsulated tablet administered in Treatment A as per protocol
  Other Names: Avelox®
Drug: Placebo Capsule — Placebo for Moxifloxacin administered in Treatment B and Treatment C

SUMMARY:
Compare the acute effect on the QT interval of MAP0004 (Dihydroergotamine Mesylate delivered by Oral Inhalation) with Moxifloxacin and Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed, executed written informed consent
2. Healthy non-smoking adult volunteers: Male or Female subjects 18 to 45 years old
3. Female subjects who are practicing adequate contraception (see section 4.4) or who are sterile
4. No known cardiac disease
5. Normal hemoglobin values
6. Normal or not clinically significant 12-lead Electrocardiogram

   * Heart rate ≥ 40 and ≤ 100 at Visit 1 vital signs assessment (resting)
   * Subjects with QTcF interval duration <430 msec for males and <450 msec for females obtained from the ECG recorder's measurements on the screening ECG taken after at least 5 minutes of quiet rest in supine position
7. Demonstrated ability to properly use the Tempo® Inhaler
8. Subject has not donated blood in the last 56 days

Exclusion Criteria:

1. Contraindication to dihydroergotamine mesylate (DHE)
2. History of hemiplegic or basilar migraine
3. Family history of long QT syndrome
4. Participation in another investigational trial during the 30 days prior to Visit 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Kori S, Kellerman DJ, Voloshko P, Haugen G. Effects of a supratherapeutic dose of investigational orally inhaled dihydroergotamine (MAP0004) on QT interval: a randomized, double-blind, active- and placebo-controlled crossover study in healthy volunteers. Clin Ther. 2012 Sep;34(9):1920-8. doi: 10.1016/j.clinthera.2012.08.001. Epub 2012 Aug 21. PMID 22917853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3-treatment, 3-period, 6-sequence crossover study. Each subject received all 3 treatments in a randomly assigned order: treatments A, B, and C, the sequences were ABC, ACB, BAC, BCA, CAB, and CBA.
Groups:
- Treatment A, Then B, Then C: Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 2.
  Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 3. Treatment C = inhaler placebo and placebo capsules at Visit 4.
- Treatment A, Then C, Then B: Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 2.
  Treatment C = inhaler placebo and placebo capsules at Visit 3. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 4.
- Treatment B, Then A, Then C: Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 2. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 3.
  Treatment C = inhaler placebo and placebo capsules at Visit 4.
- Treatment B, Then C, Then A: Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 2. Treatment C = inhaler placebo and placebo capsules at Visit 3. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 4.
- Treatment C, Then A, Then B: Treatment C = inhaler placebo and placebo capsules at Visit 2. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 3.
  Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 4.
- Treatment C, Then B, Then A: Treatment C = inhaler placebo and placebo capsules at Visit 2. Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules at Visit 3. Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet at Visit 4.
Period: Overall Study
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects enrolled in the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QTcI for MAP0004 3.0mg and Placebo at 30 Minutes
Description: The corrected QT interval, individualized (QTcI) is a measurement of the electrical impulses through the largest part of the heart muscle individualized for subject pre-dose values. A negative change is a shortening of the QTc interval, a positive change is a lengthening of the QTc interval.
Time Frame: baseline and 30 minutes
Population: Patients with data available at required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Treatment C (Placebo): Treatment C = inhaler placebo and placebo capsules.
- Treatment B (MAP0004 3.0mg): Treatment B = MAP0004 3.0mg (via inhalation) and placebo capsules.
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg)
Number analyzed (Participants) | 52 | 54
milliseconds
  Baseline | 408.8 (20.1) | 409.6 (20.9)
  Change from Baseline at 30 mins | -4.7 (6.2) | -4.6 (7.3)

2. Primary Outcome: Change From Baseline in QTcI for MAP0004 3.0mg, Placebo, and Moxifloxacin at 2 Hours
Description: as for outcome 1
Time Frame: baseline and 2 hours
Population: Patients with data available at required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Treatment C (Placebo): Treatment C = inhaler placebo and placebo capsules at Visit 3.
- Treatment A (Moxifloxacin): Treatment A = inhaler placebo and moxifloxacin 400mg encapsulated tablet.
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg) | Treatment A (Moxifloxacin)
Number analyzed (Participants) | 52 | 54 | 54
milliseconds
  Baseline | 408.8 (20.1) | 409.6 (20.9) | 408.6 (20.0)
  Change from Baseline at 2 hours | -2.3 (7.0) | -5.1 (6.7) | 9.0 (6.8)

3. Secondary Outcome: Change From Baseline in QTcF for MAP0004 3.0mg and Placebo at 30 Minutes
Description: The Fridericia corrected QT interval(QTcF) is a measurement of the electrical impulses through the largest part of the heart muscle. A negative change is a shortening of the QTc interval, a positive change is a lengthening of the QTc interval.
Time Frame: baseline and 30 minutes
Population: Patients with data available at required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg)
Number analyzed (Participants) | 52 | 54
milliseconds
  Baseline | 406.8 (18.4) | 407.7 (20.0)
  Change from Baseline at 30 mins | -5.0 (6.4) | -4.7 (6.7)

4. Secondary Outcome: Change From Baseline in QTcF for MAP0004 3.0mg, Placebo, and Moxifloxacin at 2 Hours
Description: as for outcome 3
Time Frame: baseline and 2 hours
Population: Patients with data available at required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg) | Treatment A (Moxifloxacin)
Number analyzed (Participants) | 52 | 54 | 54
milliseconds
  Baseline | 406.8 (18.4) | 407.7 (20.0) | 407.0 (18.7)
  Change from Baseline at 2 hours | -1.8 (6.9) | -3.9 (6.0) | 8.5 (6.3)

5. Secondary Outcome: Change From Baseline in Heart Rate for MAP0004 3.0mg, Placebo, and Moxifloxacin at 30 Minutes and 2 Hours
Description: The heart rate is a measure of how fast or slow the heart beats (measured in beats per minute). A negative change indicates a decrease in heart rate and a positive change indicates an increase in heart rate.
Time Frame: baseline, 30 minutes, and 2 hours
Population: Patients with data available at required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg) | Treatment A (Moxifloxacin)
Number analyzed (Participants) | 52 | 54 | 54
beats per minute (bpm)
  Baseline | 64.1 (9.1) | 64.6 (9.5) | 63.8 (9.5)
  Change from Baseline at 30 minutes | 1.0 (4.2) | -0.2 (5.8) | 2.4 (4.1)
  Change from Baseline at 2 hours | -2.1 (4.3) | -4.4 (6.7) | 0.3 (5.2)

ADVERSE EVENTS:
Description: Adverse events are presented by treatment arm, not by individual treatment (intervention) received.
Arm/Group | Treatment C (Placebo) | Treatment B (MAP0004 3.0mg) | Treatment A (Moxifloxacin)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 2/54 | 26/54 | 8/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment C (Placebo) (N=54) | Treatment B (MAP0004 3.0mg) (N=54) | Treatment A (Moxifloxacin) (N=54)
Nausea (Gastrointestinal disorders) | 0 | 15 | 2
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 5 | 4
Headache (Nervous system disorders) | 2 | 10 | 2
Paraesthesia (Nervous system disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.